CLINICAL TRIAL: NCT06323811
Title: Comparison of Free-breathing 3D Quantitative Perfusion in Patients With MINOCA, Tako-Tsubo, SCAD, Myocarditis and NSTEMI in the Acute Phase and Post Convalescence
Brief Title: Comparison of Free-breathing 3D Quantitative Perfusion in Patients With MINOCA and MINOCA-mimics
Acronym: COPE-CMR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: COPE CMR
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Myocardial Infarction With Non-Obstructive Coronary Artery; Myocarditis Acute; Takotsubo Cardiomyopathy; Spontaneous Coronary Artery Dissection; Non ST Elevation Myocardial Infarction
Keywords: MINOCA; MINOCA-mimics; CMR; 3D perfusion; advanced CMR imaging
MeSH Terms: conditions — MINOCA; Takotsubo Cardiomyopathy; Coronary Artery Dissection, Spontaneous; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: 5 groups of patients (MINOCA, myocarditis, Takotsubo cardiomyopathy, SCAD, NSTEMI) will undergo CMR with 3D perfusion in the acute setting (within 10 days after the event) and post convalescence (after 3 months)
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MINOCA (Experimental): Patients with myocardial infarction with non-obstructive coronary artery disease (MINOCA) prospectively investigated with advanced CMR
  Interventions: Diagnostic Test: CMR
- Myocarditis (Experimental): Patients with suspected myocarditis prospectively investigated with advanced CMR
  Interventions: Diagnostic Test: CMR
- Takotsubo cardiomyopathy (Experimental): Patients with suspected Takotsubo cardiomyopathy prospectively investigated with advanced CMR
  Interventions: Diagnostic Test: CMR
- Spontaneous coronary artery dissection (SCAD) (Experimental): Patients with suspected/diagnosed spontaneous coronary artery dissection prospectively investigated with advanced CMR
  Interventions: Diagnostic Test: CMR
- NSTEMI (Active Comparator): Patients with confirmed non-ST elevation myocardial infarction on coronary angiography prospectively investigated with advanced CMR
  Interventions: Diagnostic Test: CMR

INTERVENTIONS:
Diagnostic Test: CMR — Advanced CMR imaging including a novel quantitative free-breathing 3D perfusion sequence, 3D LGE imaging and a cine Dixon sequence

SUMMARY:
This clinical study examines patients presenting with acute myocardial infarction and no significant coronary artery disease on coronary angiography (MINOCA) and patients with MINOCA-mimics with advanced CMR.

The present study aims to:

* assess the microvascular function with a novel quantitative 3D myocardial perfusion imaging approach in the acute phase and post-convalescence
* refine the role and diagnostic potential of advanced quantitative CMR imaging
* assess the potential prognostic significance of microvascular dysfunction and epicardial adipose tissue on cardiovascular outcomes

Participants will undergo advanced CMR imaging in the acute setting (within 10 days after event) and post convalescence (after 3 months).

DETAILED DESCRIPTION:
Advanced CMR includes a novel free-breathing motion-informed locally low-rank quantitative 3D myocardial perfusion imaging. Perfusion imaging will be compared with 3D late gadolinium enhancement (LGE) imaging. A cine Dixon sequence is performed for the assessment of epicardial adipose tissue (EAT).

ELIGIBILITY:
Inclusion Criteria:

* acute presentation with signs/symptoms of acute coronary syndrome or myocarditis
* elevated cardiac biomarkers
* no signficant coronary artery disease on coronary angiogram or coronary CT

Exclusion Criteria:

* pacemaker/other devices or claustrophobia
* severe asthma, chronic obstructive lung or kidney disease
* acute pulmonary embolism
* arrhythmia on ECG
* moderate to severe valvular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion reserve index | within 10 days and after 3 months after index event
  comparison of microvascular function in the acute phase versus post convalescence

SECONDARY OUTCOMES:
epicardial adipose tissue (EAT) | 4 months (measured either at first or second CMR)
  the amount of epicardial adipose tissue
cardiovascular events | 5 years
  rate of cardiovascular death, myocardial infarction, recurrence of MINOCA, myocarditis, takotsubo cardiomyopathy, SCAD

CONTACTS AND LOCATIONS:
Overall Officials: Robert Manka, Prof. MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No